CLINICAL TRIAL: NCT03353103
Title: Assessment of Unstable Carotid Plaque Using PET and MR Imaging in Patient Referred to Endarterectomy: The CAROTEP Study
Brief Title: Imaging of Unstable Carotid Plaque in Patient Referred to Endarterectomy
Acronym: CAROTEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17-012
Record Dates: First submitted 2017-04-14; First posted 2017-11-27 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- symptomatic (Active Comparator)
  Interventions: Drug: Sodium fluoride F-18 PET imaging
- asymptomatic (Active Comparator)
  Interventions: Drug: Sodium fluoride F-18 PET imaging

INTERVENTIONS:
Drug: Sodium fluoride F-18 PET imaging — prior to surgical endarterectomy each patient will undergo sodium fluoride F-18 PET imaging

SUMMARY:
This study will assess unstable plaque imaging features by using high resolution MR imaging and Sodium Fluoride F-18 PET. This is a comparative study between symptomatic and asymptomatic patient referred to carotid endateriectomy, with reference to pathologic analysis of plaque components

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Health care system affiliation
* Referred to carotid endarterectomy
* Symptomatic patients:

  * Carotid stenosis between 70 and 99% (NASCET criteria)
  * TIA or minor stroke attack (RANKIN ≤ 3)
* Asymptomatic patients:

  * Carotid stenosis between 70 and 99% (NASCET criteria)
  * No symptoms
* Patient who has been informed of the study and has given his/her informed consent

Exclusion Criteria:

* Contra indication to MRI
* Renal failure (clearance < 30ml/mn)
* Patient with active inflammatory disease
* History of cancer
* Pregnancy or lactation
* Patient with carotid disease treated by fibrinolysis
* Patient under guardianship, or unable to understand the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
carotid F18-NaF uptake | baseline
  do the symptomatic patients have a higher F18-NaF uptake compared to asymptomatic patients? at pre-operative examination

SECONDARY OUTCOMES:
comparaison of F18-NaF PET and Carotid MRI | baseline
  comparaison between F18-NaF uptake and MR features of plaque instability at pre-operative examination
F18-NaF PET uptake | baseline
  comparaison between F18-NaF uptake at pre-operative imaging
histology | baseline
  comparaison between histology at post-operative histologic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided